CLINICAL TRIAL: NCT00123149
Title: An Open-Label (OL) Extension Study to Assess Safety of PROCRIT (Epoetin Alfa) in Patients With Anemia of Chronic Disease (ACD) Due to Rheumatoid Arthritis (RA)
Brief Title: Open-Label Extension Safety Study of PROCRIT in Patients With Anemia of Chronic Disease Due to Rheumatoid Arthritis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Ortho Biotech Products, L.P. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002461
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2011-07

CONDITIONS: Anemia; Rheumatoid Arthritis
Keywords: Anemia; Rheumatoid arthritis; Hemoglobin level
MeSH Terms: conditions — Anemia; Arthritis, Rheumatoid | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: Epoetin alfa

SUMMARY:
The purpose of this study is to evaluate the long-term safety profile of epoetin alfa in patients with anemia of chronic disease due to rheumatoid arthritis

DETAILED DESCRIPTION:
Epoetin alfa is an analogue of erythropoetin, a hormone secreted by kidneys known to stimulate red blood cell production. Although epoetin alfa has been known to be effective in treatment of anemia associated with chronic kidney disease, information on its effectiveness and long-term safety for treatment of anemia associated with rheumatoid arthritis is limited. This 35-week safety study is an extension of a 20-week, prospective, randomized, double-blind, placebo-controlled, multi-center study that investigates effectiveness of epoetin alfa in patients with anemia of chronic disease due to rheumatoid arthritis. The study hypothesis is that there will be no long-term safety concerns of epoetin alfa administered once every two weeks in rheumatoid arthritis patients with anemia of chronic disease. Patients will receive epoetin alfa injections (40,000 units) under their skin once every 2 weeks for up to 31 weeks. Doses may be adjusted depending on the patients' hemoglobin level up to the maximum of 60,000 units once every 2 weeks or 40,000 units once weekly.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have signed an informed consent
* Women must be postmenopausal for at least one year, surgically sterile, or practicing an effective method of birth control, or have a negative serum pregnancy test at Week 1 of the study
* Women must not be breast feeding during this study period
* Patients must have completed the double-blind (DB) study (PR03-33-055) without missing more than 4 study visits and have hemoglobin level of less than or equal to 12.9 g/dL at Week 20 of the DB study

Exclusion Criteria:

* Uncontrolled hypertension
* Elective surgery, including joint replacement, anticipated to require transfusion during the extension study period
* Thromboembolic event during the double-blind study including acute myocardial infarction, Cerebrovascular accident and/or transient ischemic attack
* Deep vein thrombosis and/or pulmonary embolism
* Uncontrolled psychiatric disease or other co-morbid disease that have developed or worsened since enrollment to the double-blind study
* Planning to be enrolled in any other clinical trial during the course of this study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Study Completion 2007-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events during the study period of up to 35 weeks; blood pressure and blood counts measured every 2 weeks up to 35 weeks. For patients who have dose increased to 40,000 units once weekly, hemoglobin levels will be monitored weekly

SECONDARY OUTCOMES:
Hemoglobin level measured every two weeks up to 35 weeks; for patients who are receiving 40,000 U QW dosing, Hb levels will be monitored weekly

CONTACTS AND LOCATIONS:
Overall Officials: Ortho Biotech Products, L.P. Clinical Trial, Study Director — Ortho Biotech Products, L.P.